CLINICAL TRIAL: NCT02687776
Title: Perioperative Copeptin: Predictive Value and Risk Stratification in Patients Undergoing Major Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2015-275
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Myocardial Injury
Keywords: Copeptin, human
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational cohort study examining the perioperative course of copeptin in patients undergoing elevated-risk surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Type of surgery for patients 1 to 30: abdominal aortic aneurysm repair, suprainguinal and infrainguinal vascular surgery, carotid surgery
* Type of surgery for patients 31 to 500: surgeries with elevated risks in general (as specified by 2014 ESC/ESA Guidelines on non-cardiac surgery:

cardiovascular assessment and management [Kristensen])

Exclusion Criteria:

* acute coronary Syndrome (ACS) at presentation (clinical assessment or documentation)
* Congestive heart failure at presentation (clinical assessment or documentation)
* Documented severe aortic stenosis (valve area <1cm2)
* Kidney dysfunction (clearance <50ml/min)
* Reduced left ventricular ejection fraction (LVEF) (<40%); if no LVEF is available, it will be assumed to be >40%
* Cancelled surgery
* Unwilling or unable to provide consent
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients >18 years undergoing major vascular surgery will be invited to participate. Specifically, patients undergoing abdominal aortic aneurysm repair, suprainguinal and infrainguinal vascular surgery, as well as carotid surgery will be included. After the first 30 patients, the population is to be expanded to elevated-risk surgeries in general.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2016-02; Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
perioperative copeptin concentrations | perioperative from induction of anesthesia to the third postoperative day
  copeptin concentrations for the perioperative time course as measured by the ThermoFisher assay at induction, at 0h, 2h, 4h, 6h, 8h, as well as on the postoperative day 1 and 3.
composite events composed of all-cause mortality and/or major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  MACCE defined as:non-fatal cardiac arrest, acute coronary syndrome (including MINS), congestive heart failure requiring hospitalization or transfer to a higher unit of care, and stroke
myocardial injury in non-cardiac surgery (MINS) | 3 postoperative days

SECONDARY OUTCOMES:
all-cause mortality | 12 months
composite events composed of all-cause mortality and/or major adverse cardiac and cerebrovascular events (MACCE) | 30 days
  MACCE: non-fatal cardiac arrest, acute coronary syndrome (including MINS), congestive heart failure requiring hospitalization or transfer to a higher unit of care, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Lurati Buse, MD, MSc, Principal Investigator — Heinrich Heine University Dusseldorf
Locations (2):
- Heinrich Heine University, Düsseldorf, Germany
- Department of Anesthesia, University of Basel Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamber F, Roth S, Bolliger D, Seeberger E, Nienhaus J, Mueller C, Lurati Buse G, Mauermann E. Perioperative copeptin: predictive value and risk stratification in patients undergoing major noncardiac surgery-a prospective observational cohort study. Can J Anaesth. 2024 Mar;71(3):330-342. doi: 10.1007/s12630-023-02677-y. Epub 2024 Jan 19. PMID 38243094
- [Derived] Kamber F, Mauermann E, Seeberger E, Guerke L, Mueller C, Bolliger D, Lurati Buse GAL. Peri-operative copeptin concentrations and their association with myocardial injury after vascular surgery: A prospective observational cohort study. Eur J Anaesthesiol. 2018 Sep;35(9):682-690. doi: 10.1097/EJA.0000000000000815. PMID 29750698